CLINICAL TRIAL: NCT02277873
Title: Two Models for Evaluate the Effect of the Proximity of the Moon on the Frequency of Births. Study on Mexican Population
Brief Title: Models for Evaluate the Proximity of the Moon on the Frequency of Births
Status: Completed | Type: Observational
Sponsor: Christian Ramos Penafiel (Other Government)
Collaborators: Instituto de Salud del Estado de Mexico (Unknown); Hospital General de Mexico (Other Government); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Sponsor-Investigator, Christian Ramos Penafiel, MD, Hospital General de Mexico
Organization: Hospital General de Mexico (Other Government)
Other Study IDs: HGM-CRP1
Record Dates: First submitted 2014-07-17; First posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Establish the Relationship Between Moon and Births
Keywords: moon; parturition; moon phases
MeSH Terms: interventions — Pregnancy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment: Defined population (pregnant women) compared on a environmental moon luminosity influence
  Interventions: Behavioral: pregnancy

INTERVENTIONS:
Behavioral: pregnancy — Observational study in order to establish relationship between moon and births
  Other Names: Statistics analysis

SUMMARY:
The purpose of this study is to establish the relationship between moon and births through two analytic models.

DETAILED DESCRIPTION:
Retrospective, descriptive and observational study. Classical model performs comparisons of births among lunar periods, lineal, cubical and exponential estimation was performed in the SPSS software and the inflection point of the curve was estimated using the formula x=[In (1/ebx)]/ebx in the Geogebra model. The significance was establish by a p value of ≤ 0.05 (95% IC).

The second analysis was performed by the difference of media between all the stages of the moon cycle as in another trials. The difference was establish by the T-student test. The difference between groups was performed by the one way ANOVA test.

This study had the review and approval from the Ethics Committee of the institution and according with Mexican regulation, and in adherence to the Helsinki declaration and International Conference for Harmonisation

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from January 2009 until June 2013

Exclusion Criteria:

* Pregnant women from any other period of time

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women from urban and rural regions from north part of Mexico city county area
Sampling Method: Non-Probability Sample
Enrollment: 25152 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
First model of analysis (Classic model) | up to 12 months
  Initial association was tempted to be done based on previous analysis described.
  The "Gibada moon" phase showed a significant difference versus Full moon and new moon, due to average birth is increased in this phase

SECONDARY OUTCOMES:
Second model of analysis. Luminosity - Births | up to 34 weeks
  For this analysis, the moon luminosity was estimated as percentage (%), as a measure of proximity between moon and the earth, and was correlated to number of births. More the percentage of light is, closest to the earth the moon is.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ramos, MD, Principal Investigator — Hospital General de Mexico
Locations (1):
- Hospital General de Cuautitlan, Cuautitlán, State of Mexico, Mexico